CLINICAL TRIAL: NCT00101816
Title: A Phase II Study of BMS-354825 in Subjects With Myeloid Blast Phase Chronic Myeloid Leukemia Resistant to or Intolerant of Imatinib Mesylate
Brief Title: Dasatinib (BMS-354825) in Subjects With Myeloid Blast Phase Chronic Myeloid Leukemia Resistant to or Intolerant of Imatinib Mesylate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-006; NCT00108719 (obsolete NCT alias)
Record Dates: First submitted 2005-01-13; First posted 2005-01-14 (Estimated); Results first posted 2010-03-02 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Myeloid Leukemia; Blast Crisis
Keywords: Myeloid blast phase Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 70 mg, twice daily, Until disease progression or intolerable toxicity, switch to the roll-over study or study closure.
  Other Names: BMS-354825; Sprycel

SUMMARY:
The purpose of this study is to see what effect an investigational drug (BMS-354825) has on subjects who are currently in the myeloid blast phase of chronic myeloid leukemia (CML) and who are either resistant to or intolerant of imatinib mesylate. Another purpose of the study is to see what side effects this drug may have on subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with myeloid blast phase chronic myeloid leukemia
* Subjects who are either resistant or intolerant of imatinib mesylate

Exclusion Criteria:

* Subjects who are eligible and willing to undergo transplantation
* Serious uncontrolled medical disorder or active infection
* Uncontrolled or significant heart problems, such as congestive heart failure, recent heart attack, etc
* Subjects receiving medications that may affect heart rhythm
* Other malignancy/cancer other than CML
* History of significant bleeding disorder unrelated to CML
* Pregnant or breastfeeding women (subjects must avoid becoming pregnant)
* Subjects received imatinib within 7 days, interferon or cytarabine within 14 days, a targeted anticancer medication within 14 days, an antineoplastic agent (other than hydroxyurea or anagrelide) within 28 days, or any other investigation medication in 28 days
* Subject is receiving medications that affect platelet function or an anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2004-12; Primary Completion 2006-08 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (62):
- United States (23):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Anaheim, California
  - Local Institution, Los Angeles, California
  - Local Institution, Stanford, California
  - Local Institution, Vallejo, California
  - Local Institution, Denver, Colorado
  - Local Institution, Jacksonville, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Kansas City, Kansas
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Detroit, Michigan
  - Local Institution, St Louis, Missouri
  - Local Institution, Hackensack, New Jersey
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Nashville, Tennessee
  - Local Institution, Houston, Texas
  - Local Institution, Seattle, Washington
- Local Institution, Adelaide, South Australia, Australia
- Local Institution, Vienna, Austria
- Belgium (2):
  - Local Institution, B-Leuven
  - Local Institution, Edegem
- Local Institution, Montreal, Quebec, Canada
- Local Institution, Aarhus, Denmark
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (3):
  - Local Institution, Hamburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Local Institution, Ramat Gan, Israel
- Italy (4):
  - Local Institution, Bologna
  - Local Institution, Napoli
  - Local Institution, Orbassano
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Trondheim, Norway
- Local Institution, Quezon City, Philippines
- Local Institution, Singapore, Singapore
- South Korea (3):
  - Local Institution, Jeollanam-Do
  - Local Institution, Kyunggi-Do
  - Local Institution, Seoul
- Sweden (4):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Local Institution, Basel, Switzerland
- Taiwan (2):
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- United Kingdom (2):
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London

REFERENCES:
- [Background] Cortes J, Rousselot P, Kim DW, Ritchie E, Hamerschlak N, Coutre S, Hochhaus A, Guilhot F, Saglio G, Apperley J, Ottmann O, Shah N, Erben P, Branford S, Agarwal P, Gollerkeri A, Baccarani M. Dasatinib induces complete hematologic and cytogenetic responses in patients with imatinib-resistant or -intolerant chronic myeloid leukemia in blast crisis. Blood. 2007 Apr 15;109(8):3207-13. doi: 10.1182/blood-2006-09-046888. Epub 2006 Dec 21. PMID 17185463
- [Background] Porkka K, Koskenvesa P, Lundan T, Rimpilainen J, Mustjoki S, Smykla R, Wild R, Luo R, Arnan M, Brethon B, Eccersley L, Hjorth-Hansen H, Hoglund M, Klamova H, Knutsen H, Parikh S, Raffoux E, Gruber F, Brito-Babapulle F, Dombret H, Duarte RF, Elonen E, Paquette R, Zwaan CM, Lee FY. Dasatinib crosses the blood-brain barrier and is an efficient therapy for central nervous system Philadelphia chromosome-positive leukemia. Blood. 2008 Aug 15;112(4):1005-12. doi: 10.1182/blood-2008-02-140665. Epub 2008 May 13. PMID 18477770

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 124 participants were enrolled in this study; 15 were never treated (11 participants did not meet inclusion criteria; 3 participants died; 1 participant failed screening).
Groups:
- Imatinib-intolerant: Defined as: i) Toxicity that was considered at least possibly related to imatinib ≤400 mg/day that led to a discontinuation of imatinib therapy ii) Ability to tolerate only <400 mg/day imatinib. A subject who tolerated 400 mg/day imatinib, but was intolerant of higher doses was not considered imatinib-intolerant. Receiving oral dasatinib at a starting dose of 70 mg twice daily (BID), with dose modifications as necessary for the management of disease progression or toxicity.
- Imatinib-resistant: Defined as any of the following: i) Subjects initially diagnosed with chronic phase chronic myeloid leukemia (CML) who progressed to myeloid phase CML while on treatment with a prescribed imatinib dose of ≥400 mg/day. ii) Subjects initially diagnosed with accelerated phase CML who progressed to myeloid phase CML while on treatment with a prescribed imatinib dose of ≥600 mg/day (or 400 to <600 mg/day if subject is intolerant of ≥600 mg/day). iii) Subjects initially diagnosed with myeloid blast phase CML who meet the criteria for myeloid phase blast crisis after at least 4 weeks of treatment prescribed at a dose of ≥600 mg/day (or 400 to <600 mg/day if subject is intolerant of ≥600 mg/day). Each of these definitions includes subjects who had no response to imatinib (primary resistance) and those who responded and subsequently progressed to myeloid blast phase (acquired resistance). Oral dasatinib 70 mg BID, with dose modifications as necessary to manage disease progression or toxicity.
Period: Overall Study
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Started | 10 | 99
Completed | 10 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 10 | 99 | 109
Age, Customized [Number; unit: participants]
  Between 21 and 45 years | 1 | 35 | 36
  Between 46 and 65 years | 7 | 46 | 53
  Between 66 and 75 years | 1 | 18 | 19
  >75 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.9) | 50.4 (14.0) | 51.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 60 | 63
  Male | 7 | 39 | 46
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 18 | 18
  Black or African American | 0 | 13 | 13
  White | 10 | 67 | 77
  Other | 0 | 1 | 1
Eastern Cooperative Oncology Group Performance Status Scale (ECOG PS) [Number; unit: Participants] — ECOG PS, a 6-item scale to assess disease progression, daily fuctioning, and appropriate treatment and prognosis. Scale: 0-5, with 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Death.
  Participants
    Score=0 | 1 | 21 | 22
    Score=1 | 6 | 39 | 45
    Score=2 | 2 | 33 | 35
    Score=3 | 0 | 2 | 2
    Score=4 | 0 | 0 | 0
    Score=5 | 0 | 0 | 0
    Not Reported | 1 | 4 | 5
Functional Assessment of Cancer Therapy-General (FACT-G) [Mean (Standard Deviation); unit: units on a scale] — FACT-G=27 questions in 4 domains: physical, social/family, emotional, & functional well-being (PWB, SWB, EWB, FWB). Score range: 0-108; higher scores=better health-related quality of life. 7 participants in the Imatinib-Intolerant group had baseline measurements; 80 participants in the Imatinib-Resistant group had baseline measurements for all 4 domains and 79 had baseline measurements for Total FACT-G scores.
  units on a scale
    Total FACT-G | 65.6 (7.1) | 69.2 (16.0) | 68.9 (15.4)
    Physical Well Being | 17.2 (3.8) | 16.4 (6.3) | 16.5 (6.1)
    Social/Family Well-Being | 20.1 (23.6) | 22.1 (4.7) | 21.9 (4.7)
    Emotional Well-Being | 15.3 (2.1) | 16.8 (5.3) | 16.7 (5.2)
    Functional Well-Being | 13.0 (4.5) | 13.9 (5.9) | 13.8 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Major and Overall Hematologic Response (MaHR and OHR)
Description: MaHR=best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL). Criteria for MaHR are specified in Outcome Measure 2. OHR=best confirmed response of MaHR or minor HR (MiHR). MiHR= <15% blasts in bone marrow and <15% blasts in peripheral blood (PB); <30% blasts + promyelocytes in bone marrow and <30% blasts + promyelocytes in PB; <20% basophils in PB; no extramedullary disease other than spleen and liver. Confirmed hematologic response=response confirmed ≥4 weeks after first documented event with no concomitant use of anagrelide or hydroxyurea.
Time Frame: Baseline (within 72 hours of therapy start); Cycle 1/Day 1; Weekly during Cycle 1 and 2; After every 2nd cycle during Cycles 3+; at end of treatment
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 10 | 99 | 109
Participants
  MaHR | 2 | 34 | 36
  OHR | 4 | 50 | 54

2. Secondary Outcome: Median Duration of Major Hematologic Response (MaHR)
Description: MaHR=best confirmed response of CHR or NEL. CHR=white blood cells ≤ institutional upper limit of normal (iULN); absolute neutrophil count (ANC) ≥1000/mm3; platelets ≥100,000/mm3; no blasts/promyelocytes in peripheral blood (PB); bone marrow blasts ≤5%; <5% myelocytes+metamyelocytes in PB; PB basophils ≤ iULN; no extramedullary involvement. NEL=WBC ≤ iULN; no blasts/promyelocytes in PB; bone marrow blasts ≤5%; <5% myelocytes+metamyelocytes in PB; PB basophils ≤ iULN; no extramedullary involvement; at least 1 of the following: ANC ≥500/mm3 & <1000/mm3; platelets ≥20,000/mm3 & <100,000/mm3.
Time Frame: as for outcome 1
Population: Participants who achieved MaHR
Measure: Median (Full Range); unit: months
Groups:
- Participants Acheiving MaHR: MaHR=best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL)
Arm/Group | Participants Acheiving MaHR
Number analyzed (Participants) | 36
months | 22.4 [1.6 to 27.3]

3. Secondary Outcome: Median Duration of Overall Hematologic Response (OHR)
Description: OHR=best confirmed response of MaHR or MiHR. MaHR=best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL). Criteria for MaHR are specified in Outcome Measure 2. Criteria for MiHR are specified in Outcome Measure 1. Maintaining a response was defined as no 2 consecutive records of non-response (ie, a single record of non-response between 2 assessments of response was not considered a loss of response).
Time Frame: as for outcome 1
Population: Participants who achieved OHR
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Participants Acheiving OHR: OHR=best confirmed response of major or minor hematologic response
Arm/Group | Participants Acheiving OHR
Number analyzed (Participants) | 54
months | 14.7 [10.0 to 22.6]

4. Secondary Outcome: Time to MaHR and OHR
Description: Median time from first dosing to date of OHR and/or MaHR in subjects who achieved OHR and MaHR. MaHR=best confirmed response of complete hematologic response (CHR) or No Evidence of Leukemia (NEL). OHR=best confirmed response of MaHR or minor hematologic response (MiHR). Criteria for MaHR are specified in Outcome Measure 2. Criteria for MiHR are specified in Outcome Measure 1.
Time Frame: as for outcome 1
Population: Participants who achieved OHR and MaHR
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Participants Acheiving OHR: OHR=best confirmed response of major or minor hematologic response (MaHR or MiHR).
Arm/Group | Participants Acheiving MaHR | Participants Acheiving OHR
Number analyzed (Participants) | 36 | 54
days | 63.5 [40.0 to 85.0] | 30.0 [29.0 to 37.0]

5. Secondary Outcome: Number of Participants With Complete, Partial, Minor, Minimal, or No Cytogenetic Response
Description: Best confirmed cytogenetic response. Determination of cytogenetic response is based on the prevalence (percentage) of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase in a bone marrow sample (aspirates/biopsies).
Time Frame: Baseline (within 4 weeks of therapy start); Every month for Cycles 1-3; Every 12 weeks for Cycles 4+; end of treatment
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 10 | 99 | 109
Participants
  Complete (0% Ph+ metaphases) | 2 | 27 | 29
  Partial (>0% to 35% Ph+ metaphases) | 0 | 8 | 8
  Minor (>35% to 65% Ph+ metaphases) | 0 | 3 | 3
  Minimal (>65% to 95% Ph+ metaphases) | 0 | 11 | 11
  No Response (>95% to 100% Ph+ metaphases) | 4 | 28 | 32
  Unable to Determine | 4 | 22 | 26

6. Secondary Outcome: Number of Participants With CHR or NEL, MiHR, or no Hematologic Response
Description: Best confirmed hematologic response. Confirmed hematologic response=response that is confirmed after at least 4 weeks with no concomitant use of anagrelide or hydroxyurea use during this interval. Criteria for complete hematologic response (CHR) or No Evidence of Leukemia (NEL) are specified in Outcome Measure 2. Criteria for minor hematologic response (MiHR) are specified in Outcome Measure 1.
Time Frame: Baseline (within 72 hours of therapy start); Cycle 1/Day 1; Weekly during Cycles 1 and 2; After every 2nd cycle for Cycles 3+; at end of treatment
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 10 | 99 | 109
Participants
  Complete | 2 | 26 | 28
  No evidence of leukemia | 0 | 8 | 8
  Minor | 2 | 16 | 18
  No response | 6 | 49 | 55

7. Secondary Outcome: Number of Participants Achieving Major Molecular Response (MMR)
Description: Number of participants who achieved an MMR at any time during the treatment period. MMR was calulated by measuring BCR-ABL transcripts in blood during treatment using quantitative reverse transcription-polymerase chain reaction (RT-PCR). BCR-ABL=the fused gene found in subjects with this type of Chronic Myeloid Leukemia (CML).
Time Frame: Baseline, every 12 weeks, and at time of Complete Cytogenetic Response (CCyR) for quantitative Polyermase Chain Reaction (qPCR) analysis
Population: treated participants with or without CCyR who were assessed for major molecular response
Measure: Number; unit: participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 3 | 45 | 48
participants
  MMR in Assessed Subjects with CCyR (n=2; n=17) | 2 | 11 | 13
  MMR in Assessed Subjects without CCyR (n=1; n=28) | 0 | 1 | 1

8. Secondary Outcome: MaHR and Major Cytogenetic Response (MCyR) Among Participants With Baseline BCR-ABL Point Mutations
Description: MaHR and MCyR in subjects with mutations at baseline, including imatinib-resistant mutations (IRM) and specific BCR-ABL mutations (SBAM). Criteria for MaHR are specified in Outcome Measure 2. MCyR=rate of complete cytogenetic responses + the rate of partial cytogenetic responses, as defined in Outcome Measure 5. BCR-ABL=the fused gene found in subjects with this type of CML. This table contains those mutations observed in at least 3 participants. The categories "1 IRM w/2-4-fold increase in resistance" and "≥1 IRM w/≥5-fold increase in resistance" refer to increase in resistance to imatinib.
Time Frame: baseline, at time of disease progression
Population: All subjects with baseline mutation data; n=the number of participants with the specified mutation. Baseline mutation data were reported for 103 of the 109 subjects (10/10 imatinib-intolerant and 93/99 imatinib-resistant). At baseline, 39 (42%) imatinib-resistant subjects and 3 imatinib-intolerant subject had imatinib-resistant mutations
Measure: Number; unit: Percentage of Participants
Groups:
- MaHR: Participants acheiving MaHR, defined as best confirmed response of Complete Hematologic Response (CHR) or No Evidence of Leukemia (NEL) of Minore Hematologic Response (MiHR)
- MCyR: Participants acheiving MCyR, defined as the rate of CCyR plus the rate of Partial Cytogenetic Response
Arm/Group | MaHR | MCyR
Number analyzed (Participants) | 103 | 103
Percentage of Participants
  Participants with IRM (n=42) | 31 | 29
  ≥1 IRM in P-loop (n=19) | 26 | 26
  ≥1 IRM in activation loop (n=8) | 38 | 13
  ≥1 IRM in other location (n=17) | 29 | 35
  ≥1 IRM w/2-4-fold increase in resistance (n=4) | 75 | 50
  ≥1 IRM w/≥5-fold increase in resistance (n=28) | 25 | 25
  SBAM [M244V] at baseline (n=3) | 33 | 33
  SBAM [G250E] at baseline (n=7) | 29 | 14
  SBAM [Y253H] at baseline (n=6) | 50 | 50
  SBAM [E255K/V] at baseline (n=5) | 0 | 20
  SBAM [T315I] at baseline (n=5) | 0 | 20
  SBAM [M351T/V] at baseline (n=3) | 67 | 67
  SBAM [F359I/V] at baseline (n=3) | 0 | 0
  SBAM [H396R] at baseline (n=4) | 25 | 0
  SBAM [F486S] at baseline (n=4) | 0 | 0

9. Secondary Outcome: Minimally Significant Changes From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G)
Description: Number of subjects with minimally significant changes from baseline in the health-related quality of life questionnaire FACT-G. FACT-G=27 questions in 4 domains: physical, social/family, emotional, & functional well-being (PWB, SWB, EWB, FWB). Score range: 0-108; higher scores=better health-related quality of life. Total Score change of 7 or more=minimal clinical important change; PWB, EWB, & FWB score change of 3 or more, & SWB score change of 2 or more=minimal clinical important change.
Time Frame: Baseline, Every 2 weeks for the first 3 cycles, following every 4-week cycle, and once at follow-up
Population: Number of participants with FACT-G assessments at baseline and at least one assessment during treatment
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 7 | 81 | 88
Participants
  Total Fact-G | 5 | 46 | 51
  Physical Well-Being | 5 | 54 | 59
  Social/Family Well-Being | 4 | 35 | 39
  Emotional Well-Being | 4 | 37 | 41
  Functional Well-Being | 3 | 42 | 45

10. Secondary Outcome: Deaths, Serious Adverse Events (SAEs), Adverse Events (AEs), AEs Leading to Discontinuation, Drug-Related AEs
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition regardless of causal relationship with treatment. SAE=any untoward medical occurrence at any dose that: results in death; is life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability; is cancer; is congenital anomaly/birth defect; results in drug dependency/abuse; is an important medical event. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: Continuously throughout study, from pre-treatment visit through end of study (due to death, unacceptable toxicity, treatment failure, etc) and follow-up period
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 10 | 99 | 109
Participants
  Death Within 30 Days | 6 | 38 | 44
  Death | 6 | 49 | 55
  SAEs | 7 | 80 | 87
  AEs | 10 | 99 | 109
  AEs Leading to Discontinuation | 3 | 39 | 42
  Drug-Related AEs | 9 | 91 | 100

11. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib - Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax was obtained from experimental observations. Using no weighting factor, the terminal log-linear phase of the concentration-time curve was identified by least-square linear regression of at least 3 data points that yielded a maximum G-criteria,which is also referred to as adjusted R-squared.
Time Frame: Collected on Days 1 and 8 at times as close as possible to the following time points (relative to drug administration): pre-dose, and following drug administration at 30 minutes, 1 hour, 1.5, 2, 3, 4, 5, 6, 8 and 10 hours.
Population: 26 participants had dense PK sampling on Day 1 and Day 8; parameters for 1 participant on Day 8 was excluded due to unreliable data. Participants with all concentration-time values < than the limit of quantitation were treated as missing for PK analysis. n= participants included in the statistical analyses of PK on Day 1 and Day 8, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 24 | 19
ng/mL | 60.34 (55.86) | 110.42 (44.31)

12. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib - Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Time Point Within the Dosing Interval of 12 h or 24 h(AUC[0-T])
Description: The AUC(0-T) was calculated using the mixed log-linear trapezoidal algorithm in Kinetica™. In the calculation of AUC(0-T), predose concentrations that were < lower limit of qualtitation were assigned a value of zero.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 24 | 19
ng∙h/mL | 161.17 (150.29) | 295.92 (169.20)

13. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib - Time to Maximum Observed Plasma Concentration (Tmax)
Description: The Tmax was obtained from experimental observations. Using no weighting factor, the terminal log-linear phase of the concentration-time curve was identified by least-square linear regression of at least 3 data points that yielded a maximum G-criteria,which is also referred to as adjusted R-squared.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 24 | 19
hours | 1.79 (1.45) [0.47 to 6.00] | 1.22 (0.97) [0.25 to 3.00]

14. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib - Plasma Half-life (T-HALF)
Description: The T-HALF was calculated as Ln2/Lz,where Lz was the absolute value of the slope of the terminal log-linear phase.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 23 | 19
hours | 3.71 (1.78) | 4.26 (2.15)

15. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib's Metabolite BMS-582691 - Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 11
Time Frame: as for outcome 11
Population: 26 participants had dense PK sampling on Day 1 & Day 8; parameters for 1 participant on Day 1 & 1 on Day 8 were excluded due to unreliable data. Participants w/all concentration-time values <than limit of quantitation were treated as missing for PK analysis. n=participants included in the statistical analyses of PK on Day 1 and Day 8, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 14 | 18
ng/mL | 2.44 (1.32) | 3.87 (1.67)

16. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib's Metabolite BMS-582691 - Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Time Point Within the Dosing Interval of 12 h (AUC[0-T])
Description: The AUC(0-T) was calculated using the mixed log-linear trapezoidal algorithm in Kinetica™. In the calculation of AUC(0-T), predose concentrations that were less than the lower limit of quantitation (LLQ) were assigned a value of zero.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Number analyzed (Participants) | 14 | 18
ng∙h/mL | 7.08 (7.80) | 13.81 (11.96)

17. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib's Metabolite BMS-582691 - Time to Maximum Observed Plasma Concentration (Tmax)
Description: as for outcome 13
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Number analyzed (Participants) | 14 | 18
hours | 1.71 (1.00) | 1.90 (1.49)

18. Secondary Outcome: Pharmacokinetics (PK) of Dasatinib and Its Metabolite BMS-582691 - Plasma Half-life (T-HALF)
Description: The T-HALF was calculated as Ln2/Lz,where Lz was the absolute value of the slope of the terminal log-linear phase.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Study Day 1 | Study Day 8
Number analyzed (Participants) | 14 | 18
hours | 4.95 (3.93) | 4.38 (3.97)

19. Secondary Outcome: Population PK of Dasatinib
Description: Population pharmacokinetic analysis was not done because it is not meaningful for this single study
Time Frame: Day 8 immediately prior to the first daily dose and between 30 minutes to 3 hours following this dose.
Measure: Number; unit: population pk
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Serious Adverse Events (participants affected / at risk) | 7/10 | 80/99
Other Adverse Events (participants affected / at risk) | 10/10 | 97/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib-intolerant (N=10) | Imatinib-resistant (N=99)
TROPONIN I (Investigations) | 0 | 1
HAEMOGLOBIN (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 1 | 1
CARDIAC ENZYMES INCREASED (Investigations) | 0 | 1
BLAST CELL COUNT INCREASED (Investigations) | 0 | 1
GRANULOCYTE COUNT DECREASED (Investigations) | 0 | 1
PLATELET AGGREGATION ABNORMAL (Investigations) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 1
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 0 | 2
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
NODAL ARRHYTHMIA (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 4
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 3
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 2
FLUSHING (Vascular disorders) | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1
HEPATOSPLENOMEGALY (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CYTOLYTIC HEPATITIS (Hepatobiliary disorders) | 0 | 1
APHASIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 3
MYELITIS (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 4
MENINGITIS NONINFECTIVE (Nervous system disorders) | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 3
ASCITES (Gastrointestinal disorders) | 0 | 1
MELAENA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 3
DIARRHOEA (Gastrointestinal disorders) | 0 | 5
GASTRITIS (Gastrointestinal disorders) | 0 | 2
STOMATITIS (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 3
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 9
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 3
SEPSIS (Infections and infestations) | 0 | 11
GANGRENE (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 0 | 5
PNEUMONIA (Infections and infestations) | 1 | 6
CELLULITIS (Infections and infestations) | 0 | 3
PHARYNGITIS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 2
BRAIN ABSCESS (Infections and infestations) | 0 | 1
LIVER ABSCESS (Infections and infestations) | 0 | 1
ANAL INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
CATHETER SEPSIS (Infections and infestations) | 0 | 1
PERIANAL ABSCESS (Infections and infestations) | 0 | 1
ASCITES INFECTION (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1
NEUTROPENIC INFECTION (Infections and infestations) | 0 | 3
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 | 1
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 3
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1
INTESTINAL STOMA (Surgical and medical procedures) | 0 | 1
STEM CELL TRANSPLANT (Surgical and medical procedures) | 0 | 1
BONE MARROW TRANSPLANT (Surgical and medical procedures) | 0 | 2
ANOREXIA (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 3
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 5
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 10
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 2
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 2
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
URTICARIA VESICULOSA (Skin and subcutaneous tissue disorders) | 0 | 1
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 0 | 1
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 | 2
FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
VERTEBRAL COLUMN MASS (Musculoskeletal and connective tissue disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 6
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 6
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 17
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 4
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PAIN (General disorders) | 0 | 1
FATIGUE (General disorders) | 0 | 1
MALAISE (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 17
ASTHENIA (General disorders) | 0 | 2
CHEST PAIN (General disorders) | 0 | 1
GENERALISED OEDEMA (General disorders) | 0 | 2
DISEASE PROGRESSION (General disorders) | 0 | 2
MUCOSAL INFLAMMATION (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
PERFORMANCE STATUS DECREASED (General disorders) | 0 | 1
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MYELOFIBROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BLAST CELL CRISIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
TUMOUR LYSIS SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
BLAST CELL PROLIFERATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 18
BLAST CRISIS IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib-intolerant (N=10) | Imatinib-resistant (N=99)
DRY EYE (Eye disorders) | 1 | 0
EYE OEDEMA (Eye disorders) | 1 | 1
EYELID OEDEMA (Eye disorders) | 1 | 4
EYE HAEMORRHAGE (Eye disorders) | 0 | 6
RETINAL HAEMORRHAGE (Eye disorders) | 1 | 1
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 | 8
CARDIAC MURMUR (Investigations) | 1 | 1
WEIGHT DECREASED (Investigations) | 5 | 25
WEIGHT INCREASED (Investigations) | 2 | 21
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 5
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 7
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 7
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
HAEMATOMA (Vascular disorders) | 1 | 7
HYPOTENSION (Vascular disorders) | 1 | 13
HYPERTENSION (Vascular disorders) | 0 | 12
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 8
INSOMNIA (Psychiatric disorders) | 2 | 13
AGITATION (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 8
DEPRESSED MOOD (Psychiatric disorders) | 2 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
GALLBLADDER ENLARGEMENT (Hepatobiliary disorders) | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 1 | 0
COMA (Nervous system disorders) | 1 | 1
APHASIA (Nervous system disorders) | 1 | 2
HEADACHE (Nervous system disorders) | 3 | 31
LETHARGY (Nervous system disorders) | 1 | 1
DIZZINESS (Nervous system disorders) | 2 | 14
CONVULSION (Nervous system disorders) | 0 | 6
SOMNOLENCE (Nervous system disorders) | 1 | 2
PARAESTHESIA (Nervous system disorders) | 0 | 5
HYPOAESTHESIA (Nervous system disorders) | 1 | 2
NAUSEA (Gastrointestinal disorders) | 3 | 34
ASCITES (Gastrointestinal disorders) | 0 | 5
VOMITING (Gastrointestinal disorders) | 6 | 37
DIARRHOEA (Gastrointestinal disorders) | 5 | 60
DYSPEPSIA (Gastrointestinal disorders) | 0 | 11
GASTRITIS (Gastrointestinal disorders) | 0 | 5
PROCTALGIA (Gastrointestinal disorders) | 1 | 4
STOMATITIS (Gastrointestinal disorders) | 3 | 14
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 21
HAEMORRHOIDS (Gastrointestinal disorders) | 2 | 7
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 22
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
LIP HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 5
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 6
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 4
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 16
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 10
RHINITIS (Infections and infestations) | 1 | 4
PNEUMONIA (Infections and infestations) | 1 | 3
ORAL HERPES (Infections and infestations) | 0 | 5
PHARYNGITIS (Infections and infestations) | 1 | 3
FOLLICULITIS (Infections and infestations) | 0 | 5
GASTROENTERITIS (Infections and infestations) | 1 | 6
NASOPHARYNGITIS (Infections and infestations) | 1 | 7
ORAL CANDIDIASIS (Infections and infestations) | 0 | 7
VAGINAL INFECTION (Infections and infestations) | 1 | 1
LOCALISED INFECTION (Infections and infestations) | 1 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 8
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 7
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
ANOREXIA (Metabolism and nutrition disorders) | 3 | 25
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 6
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 3
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 3
ANAEMIA (Blood and lymphatic system disorders) | 1 | 14
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 13
SPLENOMEGALY (Blood and lymphatic system disorders) | 1 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 17
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 6
ACNE (Skin and subcutaneous tissue disorders) | 0 | 6
RASH (Skin and subcutaneous tissue disorders) | 2 | 25
PURPURA (Skin and subcutaneous tissue disorders) | 1 | 4
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 10
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 12
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 10
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 4
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 9
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 4
SPIDER NAEVUS (Skin and subcutaneous tissue disorders) | 1 | 0
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 1 | 8
NIPPLE PAIN (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 4
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 11
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 15
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 16
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 15
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 17
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 40
RALES (Respiratory, thoracic and mediastinal disorders) | 0 | 5
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 30
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 21
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 6
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 6
NASAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 34
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 8
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 5
THROAT TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 7
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 7
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PAIN (General disorders) | 1 | 12
CHILLS (General disorders) | 0 | 12
OEDEMA (General disorders) | 1 | 9
FATIGUE (General disorders) | 3 | 34
PYREXIA (General disorders) | 8 | 62
ASTHENIA (General disorders) | 5 | 25
CHEST PAIN (General disorders) | 2 | 13
FACE OEDEMA (General disorders) | 1 | 4
HYPOTHERMIA (General disorders) | 1 | 0
PITTING OEDEMA (General disorders) | 1 | 1
LOCALISED OEDEMA (General disorders) | 3 | 4
OEDEMA PERIPHERAL (General disorders) | 3 | 35
GENERALISED OEDEMA (General disorders) | 1 | 2
MUCOSAL INFLAMMATION (General disorders) | 1 | 5
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.